CLINICAL TRIAL: NCT03636542
Title: Evaluation of Diaphragm Movement After an Interscalene Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: ANES-2018-26543
Record Dates: First submitted 2018-07-20; First posted 2018-08-17 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Phrenic Nerve Paralysis
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- liposomal bupivacaine (Experimental): These patients receive an interscalene block with liposomal bupivacaine.
  Interventions: Drug: liposomal bupivacaine
- bupivacaine (Active Comparator): These patients receive an interscalene block with bupivacaine.
  Interventions: Drug: bupivacaine

INTERVENTIONS:
Drug: liposomal bupivacaine — Experimental
  Arms: liposomal bupivacaine
Drug: bupivacaine — Active comparator
  Arms: bupivacaine

SUMMARY:
The purpose of this study is to evaluate the movement of the diaphragm after an interscalene block with liposome bupivacaine (LB) compared to interscalene block (IB) with bupivacaine. This study will evaluate if there is a possible prolonged phrenic nerve paralysis when using liposome bupivacaine in an interscalene block, using ultrasound.

DETAILED DESCRIPTION:
This study will be run concurrently with two other studies comparing bupivacaine to Liposomal Bupivacaine in shoulder surgeries. We will use already randomized patients for our randomization process. For this study in particular we will use an ultrasound machine to scan the diaphragm of any patient who had an Interscalene Block for Total Shoulder Arthroplasy or Rotator Cuff Repair. Patients are to be scanned in an upright sitting position and scanned from a low intercostal or subcostal approach using the liver or spleen as an acoustic window. M Mode will be applied and the range of diaphragmatic movement from the resting expiratory position to deep inspiration (sigh test) will be recorded as was the range of diaphragmatic movement from resting expiratory position when quickly inspiring through the nose (sniff test). The blocks will be done regardless of the study as they are standard of care for pain control. The only intervention is ultrasound examination of the patient's diaphragm at baseline, 3 hours post block in recovery room and on post-operative day 1, and basic spirometry to record FEV1 and FVC via a portable spirometer at the same time points. If patients did stay in hospital on postoperative day 2 we would also evaluate their diaphragm function.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 years and older who are scheduled for shoulder surgery with interscalene block and remain in the hospital for more than 24 hours that are being randomized into a bupivacaine versus liposomal bupivacaine interscalene block study.

Exclusion Criteria:

* Non English speaking patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason habeck, MD, Principal Investigator — University of Minnesota
Locations (1):
- Univeristy of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Started | 12 | 14
Completed | 10 | 12
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Bupivacaine | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 6 | 10 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Diaphragm Excursion With Sigh
Description: Evaluation of diaphragm excursion (movement in cm) from rest to sigh in a sitting position.
Time Frame: change from baseline to 24 hours after block
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 12 | 10
cm | 4.2 [1.6 to 5.0] | 2.9 [1.7 to 3.5]

2. Secondary Outcome: Diaphragm Excursion With Quick Inspiratory Breath
Description: Evaluation of diaphragm excursion (movement in cm) from rest to a quick inspiratory breath.
Time Frame: change from baseline to 24 hours after block
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 9 | 12
cm | 1.8 [1.3 to 2.9] | 1.2 [0.7 to 2.3]

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Evaluation of FEV1 via spirometry.
Time Frame: change from baseline to 24 hours after block
Measure: Median (Inter-Quartile Range); unit: liters
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 10 | 12
liters | 2.7 [1.9 to 3.2] | 1.8 [1.7 to 2.1]

4. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Evaluation of FVC via spirometry.
Time Frame: change from baseline to 24 hours after block
Measure: Median (Inter-Quartile Range); unit: liters
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 10 | 12
liters | 3.2 [2.3 to 3.5] | 2.0 [1.8 to 2.3]

5. Secondary Outcome: FEV1/FVC
Description: Evaluation of FEV1/FVC percent via spirometry.
Time Frame: change from baseline to 24 hours after block
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Number analyzed (Participants) | 10 | 12
percent | 86 [86.2 to 97.3] | 89.5 [82.3 to 93.0]

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Liposomal Bupivacaine | Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT03636542/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT03636542/ICF_001.pdf